CLINICAL TRIAL: NCT01740791
Title: Phase 1b, Randomized, Double-Blind, Multiple-Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of GS-5816 in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Velpatasvir in Participants With Chronic HCV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-281-0102
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Chronic Hepatitis C Virus
Keywords: Hepatitis C; HCV; Genotype 1; Genotype 2; Genotype 3; Genotype 4; Genotype 5; Genotype 6; Liver Disease
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Diseases | interventions — velpatasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Velpatasvir 5 mg (GT 1a) (Experimental): Participants with genotype (GT) 1a HCV infection will receive velpatasvir 5 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 25 mg (GT 1a) (Experimental): Participants with GT 1a HCV infection will receive velpatasvir 25 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 50 mg (GT 1a) (Experimental): Participants with GT 1a HCV infection will receive velpatasvir 50 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 100 mg (GT 1a) (Experimental): Participants with GT 1a HCV infection will receive velpatasvir 100 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 150 mg (GT 1a) (Experimental): Participants with GT 1a HCV infection will receive velpatasvir 150 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 150 mg (GT 1b) (Experimental): Participants with GT 1b HCV infection will receive velpatasvir 150 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 150 mg (GT 2) (Experimental): Participants with GT 2 HCV infection will receive velpatasvir 150 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 25 mg (GT 3) (Experimental): Participants with GT 3 HCV infection will receive velpatasvir 25 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 50 mg (GT 3) (Experimental): Participants with GT 3 HCV infection will receive velpatasvir 50 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 150 mg (GT 3) (Experimental): Participants with GT 3 HCV infection will receive velpatasvir 150 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir 150 mg (GT 4) (Experimental): Participants with GT 4 HCV infection will receive velpatasvir 150 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo
- Velpatasvir up to 400 mg (GT 2) (Experimental): Participants with GT 2 HCV infection will receive velpatasvir up to 400 mg or placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Velpatasvir; Drug: Placebo

INTERVENTIONS:
Drug: Velpatasvir — Tablets administered orally
  Other Names: GS-5816
Drug: Placebo — Tablets administered orally

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, and antiviral activity of velpatasvir (formerly GS-5816) in HCV treatment naive participants with genotypes 1-6.

ELIGIBILITY:
Key Inclusion Criteria:

* HCV treatment-naive adult participants (18-65 years of age) with chronic HCV infection and plasma HCV RNA ≥ 5 log10 IU/mL at screening
* Agree to use protocol defined precautions against pregnancy

Key Exclusion Criteria:

* Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
* Evidence of cirrhosis
* Evidence of current drug abuse
* Screening laboratory results outside the protocol specified requirements

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2013-03-15 (Actual); Study Completion 2014-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (10):
- United States (9):
  - West Coast Clinical Trials, LLC, Costa Mesa, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - CRI Worldwide, LLC, Marlton, New Jersey
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - New Orleans Center for Clinical Research-Knoxville, Knoxville, Tennessee
  - Alamo Medical Research, San Antonio, Texas
  - Charles River Clinical Services Northwest, Inc., Tacoma, Washington
- Fundacion De Investigacion De Diego, San Juan, Puerto Rico

REFERENCES:
- [Result] Hebner C, Gontcharova V, Chodavarapu RK, Rodriguez-Torres M, Lawitz E, Yang C, et al. Deep Sequencing of HCV NS5A From a 3-Day Study of GS-5816 Monotherapy Confirms the Potency of GS-5816 Against Pre-Existing Genotype 1-3 NS5A Resistance-Associated Variants [Abstract 470]. The Liver Meeting The 64th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD); 2013 November 1-5; Washington, D.C.
- [Result] Lawitz E, Glass SJ, Gruener D, Freilich B, Hill JM, Link JO, et al. GS-5816, a Once-Daily NS5A Inhibitor, Demonstrates Potent Antiviral Activity in Patients with Genotype 1, 2, 3, or 4 HCV Infection in a 3-Day Monotherapy Study [Abstract 1082]. The Liver Meeting The 64th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD); 2013 November 1-5; Washington, D.C.
- [Derived] Lawitz EJ, Dvory-Sobol H, Doehle BP, Worth AS, McNally J, Brainard DM, Link JO, Miller MD, Mo H. Clinical Resistance to Velpatasvir (GS-5816), a Novel Pan-Genotypic Inhibitor of the Hepatitis C Virus NS5A Protein. Antimicrob Agents Chemother. 2016 Aug 22;60(9):5368-78. doi: 10.1128/AAC.00763-16. Print 2016 Sep. PMID 27353271
- [Derived] Lawitz E, Freilich B, Link J, German P, Mo H, Han L, Brainard DM, McNally J, Marbury T, Rodriguez-Torres M. A phase 1, randomized, dose-ranging study of GS-5816, a once-daily NS5A inhibitor, in patients with genotype 1-4 hepatitis C virus. J Viral Hepat. 2015 Dec;22(12):1011-9. doi: 10.1111/jvh.12435. Epub 2015 Jul 16. PMID 26183611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 06 November 2012. The last study visit occurred on 24 January 2014.
Pre-assignment Details: 163 participants were screened. Participants were not enrolled in 'Velpatasvir up to 400 mg genotype (GT) 2' group.
Groups:
- Placebo: Participants with HCV infection received placebo once daily for 3 days under fasted conditions.
- Velpatasvir 5 mg: Participants with HCV infection received velpatasvir 5 mg once daily for 3 days under fasted conditions.
- Velpatasvir 25 mg: Participants with HCV infection received velpatasvir 25 mg once daily for 3 days under fasted conditions.
- Velpatasvir 50 mg: Participants with HCV infection received velpatasvir 50 mg once daily for 3 days under fasted conditions.
- Velpatasvir 100 mg: Participants with HCV infection received velpatasvir 100 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg: Participants with HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
Period: Overall Study
Arm/Group | Placebo | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Started | 22 | 7 | 17 | 14 | 9 | 34
Completed | 10 | 4 | 11 | 7 | 6 | 23
Not Completed | 12 | 3 | 6 | 7 | 3 | 11
Not completed — Randomized but never treated | 5 | 3 | 2 | 2 | 1 | 3
Not completed — Lost to Follow-up | 2 | 0 | 2 | 3 | 2 | 3
Not completed — Withdrew Consent | 4 | 0 | 1 | 2 | 0 | 3
Not completed — Investigator's discretion | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug (velpatasvir or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg | Total
Number analyzed (Participants) | 17 | 4 | 15 | 12 | 8 | 31 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.46) | 44.8 (15.65) | 45.1 (11.56) | 46.9 (10.13) | 47.0 (8.40) | 49.2 (9.12) | 47.3 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 2 | 2 | 8 | 19
  Male | 14 | 3 | 12 | 10 | 6 | 23 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 0 | 5 | 4 | 2 | 10 | 27
  White | 11 | 4 | 10 | 7 | 6 | 21 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 3 | 6 | 2 | 8 | 28
  Not Hispanic or Latino | 9 | 3 | 12 | 6 | 6 | 23 | 59
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.52 (0.517) | 6.64 (0.312) | 6.32 (0.826) | 6.39 (0.558) | 6.46 (0.479) | 6.41 (0.603) | 6.43 (0.597)
HCV Genotype [Count of Participants; unit: Participants]
  1a | 10 | 4 | 8 | 8 | 8 | 7 | 45
  1b | 2 | 0 | 0 | 0 | 0 | 8 | 10
  2b | 2 | 0 | 0 | 0 | 0 | 8 | 10
  3 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  3a | 3 | 0 | 6 | 4 | 0 | 6 | 19
  4 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  4a/4c/4d | 0 | 0 | 0 | 0 | 0 | 1 | 1
IL28B Genotype [Count of Participants; unit: Participants]
  C/C | 7 | 2 | 5 | 5 | 2 | 5 | 26
  C/T | 5 | 2 | 8 | 5 | 6 | 18 | 44
  T/T | 5 | 0 | 2 | 2 | 0 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events
Description: Treatment-emergent adverse events were defined as any new or worsening adverse event that began on or after the date of the first dose of study drug until the Day 17 study visit date + 2 (Day 19 if Day 17 visit missing).
Time Frame: First dose date up to Day 17 + 2 (Day 19 if Day 17 visit missing)
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug (velpatasvir or placebo). Data were summarized by velpatasvir or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 17 | 4 | 15 | 12 | 8 | 31
percentage of participants | 17.6 | 25.0 | 26.7 | 8.3 | 37.5 | 29.0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from baseline at any postbaseline visit up to the Day 17 visit date + 2 days (or Day 19 if Day 17 visit was missing). The criteria used to grade laboratory results were as follows: Grade 1 (mild), Grade 2 (moderate), or Grade 3 (severe). Graded laboratory abnormalities were defined using the grading scheme defined in protocol (Gilead Sciences, Inc. Grading Scale for Severity of Adverse Events and Laboratory Abnormalities) for analysis purpose.
Time Frame: First dose date up to Day 17 + 2 (Day 19 if Day 17 visit missing)
Population: Participants in the Safety Analysis Set were analyzed. Data were summarized by dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 17 | 4 | 15 | 12 | 8 | 31
percentage of participants
  Grade 1 | 41.2 | 25.0 | 40.0 | 58.3 | 62.5 | 33.3
  Grade 2 | 17.6 | 0 | 33.3 | 8.3 | 25.0 | 33.3
  Grade 3 | 11.8 | 0 | 13.3 | 16.7 | 0 | 6.7

3. Primary Outcome: Antiviral Activity of Velpatasvir as Measured by Change in Plasma HCV RNA From Baseline
Description: Participants who were genotyped incorrectly but received appropriate treatment for that genotype were included in that treatment group for the efficacy analysis. Data were summarized by treatment and placebo.
Time Frame: Baseline; Days 4, 5, 6, 7, 8, 10, and 17
Population: Participants in the Efficacy Analysis Set (all randomized participants with appropriate genotype who received at least one dose of the study drug (velpatasvir or placebo) and with at least one on-treatment HCV RNA assessment) with available data were analyzed. Data were summarized by treatment (velpatasvir dose/HCV genotype) and placebo.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Velpatasvir 5 mg (GT 1a): Participants with genotype (GT) 1a HCV infection received velpatasvir 5 mg once daily for 3 days under fasted conditions.
- Velpatasvir 25 mg (GT 1a): Participants with GT 1a HCV infection received velpatasvir 25 mg once daily for 3 days under fasted conditions.
- Velpatasvir 50 mg (GT 1a): Participants with GT 1a HCV infection received velpatasvir 50 mg once daily for 3 days under fasted conditions.
- Velpatasvir 100 mg (GT 1a): Participants with GT 1a HCV infection received velpatasvir 100 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 1a): Participants with GT 1a HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 1b): Participants with GT 1b HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 2): Participants with GT 2 HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 25 mg (GT 3): Participants with GT 3 HCV infection received velpatasvir 25 mg once daily for 3 days under fasted conditions.
- Velpatasvir 50 mg (GT 3): Participants with GT 3 HCV infection received velpatasvir 50 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 3): Participants with GT 3 HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 4): Participants with GT 4 HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
Arm/Group | Placebo | Velpatasvir 5 mg (GT 1a) | Velpatasvir 25 mg (GT 1a) | Velpatasvir 50 mg (GT 1a) | Velpatasvir 100 mg (GT 1a) | Velpatasvir 150 mg (GT 1a) | Velpatasvir 150 mg (GT 1b) | Velpatasvir 150 mg (GT 2) | Velpatasvir 25 mg (GT 3) | Velpatasvir 50 mg (GT 3) | Velpatasvir 150 mg (GT 3) | Velpatasvir 150 mg (GT 4)
Number analyzed (Participants) | 17 | 4 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 4 | 6 | 2
log10 IU/mL
  Change at Day 4: number analyzed (Participants) | 17 | 4 | 8 | 8 | 8 | 7 | 7 | 8 | 6 | 4 | 6 | 2
  Change at Day 4 | -0.005 (0.3343) | -3.104 (0.7348) | -3.638 (0.4350) | -3.338 (1.3088) | -3.154 (1.0089) | -3.648 (0.9270) | -3.848 (0.4834) | -4.044 (0.3671) | -2.796 (1.4313) | -2.382 (1.5028) | -2.834 (0.7608) | -3.269 (0.6080)
  Change at Day 5: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 7 | 7 | 6 | 6 | 4 | 6 | 2
  Change at Day 5 | -0.018 (0.2346) | -1.998 (0.8305) | -3.538 (0.7566) | -3.123 (1.5009) | -3.060 (1.1098) | -3.636 (1.0023) | -3.955 (0.3519) | -4.148 (0.5841) | -2.617 (1.3034) | -2.130 (1.4385) | -2.259 (1.1488) | -2.827 (0.5506)
  Change at Day 6: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 6 | 7 | 8 | 6 | 4 | 6 | 2
  Change at Day 6 | -0.037 (0.2119) | -1.244 (0.6135) | -3.140 (0.9786) | -2.704 (1.5100) | -2.713 (1.1206) | -3.221 (1.2323) | -4.021 (0.3681) | -4.109 (0.6408) | -2.193 (1.1060) | -1.737 (1.3854) | -1.869 (1.3270) | -2.243 (0.5919)
  Change at Day 7: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 5 | 7 | 8 | 6 | 4 | 6 | 2
  Change at Day 7 | -0.003 (0.1923) | -1.031 (0.6112) | -2.424 (0.7292) | -2.184 (1.5527) | -2.273 (1.1753) | -2.481 (1.3542) | -4.205 (0.4393) | -3.850 (0.9630) | -1.586 (1.0710) | -1.742 (1.3842) | -1.380 (1.6686) | -1.892 (1.0143)
  Change at Day 8: number analyzed (Participants) | 16 | 4 | 8 | 8 | 8 | 7 | 7 | 8 | 6 | 4 | 6 | 2
  Change at Day 8 | 0.027 (0.2740) | -0.941 (0.5345) | -2.074 (0.7701) | -1.702 (1.6152) | -1.780 (0.9987) | -2.544 (1.5460) | -4.026 (0.3155) | -3.559 (0.9866) | -1.025 (1.1864) | -1.542 (1.0593) | -1.062 (1.5998) | -1.478 (1.1542)
  Change at Day 10: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 6 | 7 | 8 | 6 | 4 | 6 | 2
  Change at Day 10 | 0.142 (0.3813) | -0.679 (0.4352) | -1.304 (1.0374) | -1.472 (1.4315) | -1.143 (1.2137) | -2.032 (1.4388) | -3.348 (0.6201) | -2.918 (1.1566) | -0.844 (0.6967) | -1.051 (1.4338) | -1.198 (1.0991) | -0.494 (0.8933)
  Change at Day 17: number analyzed (Participants) | 16 | 4 | 8 | 7 | 8 | 7 | 7 | 8 | 6 | 3 | 6 | 2
  Change at Day 17 | -0.025 (0.2719) | -0.135 (0.3747) | -0.223 (0.4236) | -1.110 (1.3584) | -0.801 (0.7679) | -0.879 (0.9231) | -1.532 (1.2059) | -0.886 (1.3190) | -0.672 (0.5003) | -0.085 (0.6910) | -0.225 (0.4210) | -0.351 (0.5914)

4. Secondary Outcome: Absolute HCV RNA Level
Time Frame: Baseline; Days 4, 5, 6, 7, 8, 10, and 17
Population: Participants in the Efficacy Analysis Set with available data were analyzed. Data were summarized by treatment (velpatasvir dose/HCV genotype) and placebo.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Velpatasvir 5 mg (GT 1a): Participants with GT 1a HCV infection received velpatasvir 5 mg once daily for 3 days under fasted conditions.
Arm/Group | Placebo | Velpatasvir 5 mg (GT 1a) | Velpatasvir 25 mg (GT 1a) | Velpatasvir 50 mg (GT 1a) | Velpatasvir 100 mg (GT 1a) | Velpatasvir 150 mg (GT 1a) | Velpatasvir 150 mg (GT 1b) | Velpatasvir 150 mg (GT 2) | Velpatasvir 25 mg (GT 3) | Velpatasvir 50 mg (GT 3) | Velpatasvir 150 mg (GT 3) | Velpatasvir 150 mg (GT 4)
Number analyzed (Participants) | 17 | 4 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 4 | 6 | 2
log10 IU/mL
  Baseline | 6.523 (0.5173) | 6.639 (0.3123) | 6.461 (0.6623) | 6.459 (0.5726) | 6.458 (0.4785) | 6.335 (0.5710) | 6.379 (0.4187) | 6.753 (0.5857) | 6.150 (1.0108) | 6.240 (0.5796) | 6.318 (0.8151) | 5.734 (0.2345)
  Day 4: number analyzed (Participants) | 17 | 4 | 8 | 8 | 8 | 7 | 7 | 8 | 6 | 4 | 6 | 2
  Day 4 | 6.518 (0.4840) | 3.535 (0.7588) | 2.823 (0.7866) | 3.121 (1.6969) | 3.304 (1.2823) | 2.687 (0.8776) | 2.574 (0.3526) | 2.708 (0.5823) | 3.151 (2.0090) | 3.858 (1.9120) | 3.484 (0.6784) | 2.465 (0.8425)
  Day 5: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 7 | 7 | 6 | 6 | 4 | 6 | 2
  Day 5 | 6.512 (0.5715) | 4.642 (0.9016) | 2.922 (1.0852) | 3.336 (1.8716) | 3.398 (1.3325) | 2.699 (1.0083) | 2.466 (0.3511) | 2.681 (0.3893) | 3.329 (1.8305) | 4.110 (1.8964) | 4.059 (1.0186) | 2.907 (0.7850)
  Day 6: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 6 | 7 | 8 | 6 | 4 | 6 | 2
  Day 6 | 6.493 (0.5373) | 5.395 (0.6898) | 3.321 (1.3322) | 3.755 (1.9323) | 3.745 (1.3213) | 3.104 (1.2373) | 2.400 (0.3365) | 2.644 (0.6568) | 3.753 (1.6214) | 4.503 (1.9383) | 4.450 (1.1943) | 3.491 (0.8264)
  Day 7: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 5 | 7 | 8 | 6 | 4 | 6 | 2
  Day 7 | 6.527 (0.6190) | 5.608 (0.6929) | 4.036 (1.1305) | 4.275 (1.9196) | 4.185 (1.4107) | 3.862 (1.4141) | 2.217 (0.5807) | 2.903 (0.7639) | 4.361 (1.4130) | 4.498 (1.9226) | 4.938 (1.4707) | 3.842 (1.2488)
  Day 8: number analyzed (Participants) | 16 | 4 | 8 | 8 | 8 | 7 | 7 | 8 | 6 | 4 | 6 | 2
  Day 8 | 6.555 (0.4880) | 5.699 (0.6305) | 4.387 (1.1089) | 4.756 (1.9494) | 4.678 (1.3233) | 3.791 (1.5984) | 2.396 (0.6092) | 3.194 (0.8402) | 4.922 (1.3395) | 4.698 (1.6047) | 5.256 (1.3141) | 4.256 (1.3887)
  Day 10: number analyzed (Participants) | 15 | 4 | 8 | 8 | 8 | 6 | 7 | 8 | 6 | 4 | 6 | 2
  Day 10 | 6.659 (0.4583) | 5.960 (0.6104) | 5.156 (1.3456) | 4.986 (1.7558) | 5.315 (1.5130) | 4.319 (1.6357) | 3.074 (0.8660) | 3.834 (1.1710) | 5.103 (1.1273) | 5.190 (2.0061) | 5.120 (0.6140) | 5.240 (1.1278)
  Day 17: number analyzed (Participants) | 16 | 4 | 8 | 7 | 8 | 7 | 7 | 8 | 6 | 4 | 6 | 2
  Day 17 | 6.503 (0.5432) | 6.505 (0.5615) | 6.237 (0.6709) | 5.468 (1.6269) | 5.657 (1.0148) | 5.455 (1.2889) | 4.890 (1.5438) | 5.867 (1.5443) | 5.275 (1.1421) | 6.007 (0.9524) | 6.093 (0.6451) | 5.383 (0.8259)

5. Secondary Outcome: Number of Participants Achieving Reductions From Baseline in HCV RNA
Description: Categorical declines from baseline were summarized by the number of participants with a < 1, ≥ 1 to < 2, ≥ 2 to < 3, or ≥ 3 log10 IU/mL decrease in HCV RNA from baseline by treatment (velpatasvir dose/HCV genotype) and placebo at each collection time point through Day 17.
Time Frame: Baseline; Days 4, 5, 6, 7, 8, 10, and 17
Population: Participants in the Efficacy Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Velpatasvir 5 mg (GT 1a) | Velpatasvir 25 mg (GT 1a) | Velpatasvir 50 mg (GT 1a) | Velpatasvir 100 mg (GT 1a) | Velpatasvir 150 mg (GT 1a) | Velpatasvir 150 mg (GT 1b) | Velpatasvir 150 mg (GT 2) | Velpatasvir 25 mg (GT 3) | Velpatasvir 50 mg (GT 3) | Velpatasvir 150 mg (GT 3) | Velpatasvir 150 mg (GT 4)
Number analyzed (Participants) | 17 | 4 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 4 | 6 | 2
Participants
  Day 4: Missing HCV RNA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Day 4: < 1 log10 IU/mL decrease in HCV RNA | 17 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Day 4: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Day 4: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 1 | 3 | 1
  Day 4: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 3 | 7 | 5 | 4 | 5 | 7 | 8 | 4 | 2 | 2 | 1
  Day 5: Missing HCV RNA | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
  Day 5: < 1 log10 IU/mL decrease in HCV RNA | 15 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Day 5: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 5: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 2 | 2 | 1
  Day 5: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 7 | 5 | 4 | 5 | 7 | 6 | 3 | 1 | 2 | 1
  Day 6: Missing HCV RNA | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Day 6: < 1 log10 IU/mL decrease in HCV RNA | 15 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
  Day 6: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 3 | 1 | 2 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 1
  Day 6: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1
  Day 6: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 7 | 5 | 4 | 4 | 7 | 7 | 2 | 0 | 2 | 0
  Day 7: Missing HCV RNA | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
  Day 7: < 1 log10 IU/mL decrease in HCV RNA | 15 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 2 | 1 | 3 | 0
  Day 7: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1
  Day 7: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 5 | 3 | 3 | 0 | 0 | 3 | 3 | 2 | 0 | 1
  Day 7: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 2 | 2 | 3 | 3 | 7 | 5 | 0 | 0 | 2 | 0
  Day 8: Missing HCV RNA | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Day 8: < 1 log10 IU/mL decrease in HCV RNA | 16 | 2 | 1 | 3 | 2 | 2 | 0 | 0 | 3 | 1 | 4 | 1
  Day 8: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Day 8: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 5 | 1 | 3 | 2 | 0 | 3 | 2 | 2 | 2 | 1
  Day 8: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 2 | 1 | 3 | 7 | 5 | 0 | 0 | 0 | 0
  Day 10: Missing HCV RNA | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Day 10: < 1 log10 IU/mL decrease in HCV RNA | 15 | 3 | 3 | 4 | 3 | 1 | 0 | 0 | 4 | 2 | 3 | 1
  Day 10: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 1 | 4 | 2 | 3 | 2 | 0 | 2 | 2 | 0 | 1 | 1
  Day 10: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 2 | 0 | 2 | 2 | 0
  Day 10: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 4 | 0 | 0 | 0 | 0
  Day 17: Missing HCV RNA | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Day 17: < 1 log10 IU/mL decrease in HCV RNA | 16 | 4 | 8 | 5 | 5 | 6 | 3 | 6 | 5 | 3 | 6 | 2
  Day 17: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Day 17: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Day 17: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Have HCV RNA < Lower Limit of Quantitation (LLOQ) Detected
Description: The lower limit of quantitation (LLOQ) detection for HCV RNA levels was 25 IU/mL. HCV detected means calculated HCV RNA level is below LLOQ of the assay.
Time Frame: Days 4, 5, 6, 7, and 8
Population: Participants in the Efficacy Analysis Set were analyzed. Data were summarized by treatment (velpatasvir dose/HCV genotype) and placebo.
Measure: Number; unit: participants
Arm/Group | Placebo | Velpatasvir 5 mg (GT 1a) | Velpatasvir 25 mg (GT 1a) | Velpatasvir 50 mg (GT 1a) | Velpatasvir 100 mg (GT 1a) | Velpatasvir 150 mg (GT 1a) | Velpatasvir 150 mg (GT 1b) | Velpatasvir 150 mg (GT 2) | Velpatasvir 25 mg (GT 3) | Velpatasvir 50 mg (GT 3) | Velpatasvir 150 mg (GT 3) | Velpatasvir 150 mg (GT 4)
Number analyzed (Participants) | 17 | 4 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 4 | 6 | 2
participants
  Day 4 < LLOQ detected | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Day 5 < LLOQ detected | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Day 6 < LLOQ detected | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7 < LLOQ detected | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 < LLOQ detected | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Plasma HCV RNA Levels by Treatment and IL28B Genotype
Time Frame: Days 4, 5, 6, 7, 8, 10, and 17
Population: Participants in the Efficacy Analysis Set with available data were analyzed. Data are were summarized by treatment (velpatasvir dose/HCV genotype and placebo) and IL28B genotype (CC and non-CC). Due to the small number of participants in each treatment group, no conclusions can be made on the effect of IL28B genotype on HCV RNA decline.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Placebo (IL28B Genotype CC); Placebo (IL28B Genotype Non-CC): Participants with HCV infection received placebo once daily for 3 days under fasted conditions.
- Velpatasvir 5 mg (GT 1a) (IL28B Genotype CC); Velpatasvir 5 mg (GT 1a) (IL28B Genotype Non-CC): Participants with GT 1a HCV infection received velpatasvir 5 mg once daily for 3 days under fasted conditions.
- Velpatasvir 25 mg (GT 1a) (IL28B Genotype CC); Velpatasvir 25 mg (GT 1a) (IL28B Genotype Non-CC): Participants with GT 1a HCV infection received velpatasvir 25 mg once daily for 3 days under fasted conditions.
- Velpatasvir 50 mg (GT 1a) (IL28B Genotype CC); Velpatasvir 50 mg (GT 1a) (IL28B Genotype Non-CC): Participants with GT 1a HCV infection received velpatasvir 50 mg once daily for 3 days under fasted conditions.
- Velpatasvir 100 mg (GT 1a) (IL28B Genotype CC); Velpatasvir 100 mg (GT 1a) (IL28B Genotype Non-CC): Participants with GT 1a HCV infection received velpatasvir 100 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 1a) (IL28B Genotype CC); Velpatasvir 150 mg (GT 1a) (IL28B Genotype Non-CC): Participants with GT 1a HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 1b) (IL28B Genotype CC); Velpatasvir 150 mg (GT 1b) (IL28B Genotype Non-CC): Participants with GT 1b HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 2) (IL28B Genotype CC); Velpatasvir 150 mg (GT 2) (IL28B Genotype Non-CC): Participants with GT 2 HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 25 mg (GT 3) (IL28B Genotype CC); Velpatasvir 25 mg (GT 3) (IL28B Genotype Non-CC): Participants with GT 3 HCV infection received velpatasvir 25 mg once daily for 3 days under fasted conditions.
- Velpatasvir 50 mg (GT 3) (IL28B Genotype CC); Velpatasvir 50 mg (GT 3) (IL28B Genotype Non-CC): Participants with GT 3 HCV infection received velpatasvir 50 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 3) (IL28B Genotype CC); Velpatasvir 150 mg (GT 3) (IL28B Genotype Non-CC): Participants with GT 3 HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
- Velpatasvir 150 mg (GT 4) (IL28B Genotype CC); Velpatasvir 150 mg (GT 4) (IL28B Genotype Non-CC): Participants with GT 4 HCV infection received velpatasvir 150 mg once daily for 3 days under fasted conditions.
Arm/Group | Placebo (IL28B Genotype CC) | Velpatasvir 5 mg (GT 1a) (IL28B Genotype CC) | Velpatasvir 25 mg (GT 1a) (IL28B Genotype CC) | Velpatasvir 50 mg (GT 1a) (IL28B Genotype CC) | Velpatasvir 100 mg (GT 1a) (IL28B Genotype CC) | Velpatasvir 150 mg (GT 1a) (IL28B Genotype CC) | Velpatasvir 150 mg (GT 1b) (IL28B Genotype CC) | Velpatasvir 150 mg (GT 2) (IL28B Genotype CC) | Velpatasvir 25 mg (GT 3) (IL28B Genotype CC) | Velpatasvir 50 mg (GT 3) (IL28B Genotype CC) | Velpatasvir 150 mg (GT 3) (IL28B Genotype CC) | Velpatasvir 150 mg (GT 4) (IL28B Genotype CC) | Placebo (IL28B Genotype Non-CC) | Velpatasvir 5 mg (GT 1a) (IL28B Genotype Non-CC) | Velpatasvir 25 mg (GT 1a) (IL28B Genotype Non-CC) | Velpatasvir 50 mg (GT 1a) (IL28B Genotype Non-CC) | Velpatasvir 100 mg (GT 1a) (IL28B Genotype Non-CC) | Velpatasvir 150 mg (GT 1a) (IL28B Genotype Non-CC) | Velpatasvir 150 mg (GT 1b) (IL28B Genotype Non-CC) | Velpatasvir 150 mg (GT 2) (IL28B Genotype Non-CC) | Velpatasvir 25 mg (GT 3) (IL28B Genotype Non-CC) | Velpatasvir 50 mg (GT 3) (IL28B Genotype Non-CC) | Velpatasvir 150 mg (GT 3) (IL28B Genotype Non-CC) | Velpatasvir 150 mg (GT 4) (IL28B Genotype Non-CC)
Number analyzed (Participants) | 7 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 2 | 3 | 1 | 0 | 10 | 2 | 5 | 6 | 6 | 7 | 7 | 5 | 5 | 1 | 5 | 2
log10 IU/mL
  Day 4: number analyzed (Participants) | 7 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 1 | 0 | 10 | 2 | 5 | 6 | 6 | 7 | 6 | 5 | 5 | 1 | 5 | 2
  Day 4 | 6.473 (0.4869) | 3.410 (0.4007) | 2.603 (0.5255) | 1.762 (0.5394) | 2.891 (0.4237) |  | 2.539 | 2.758 (0.3416) | 2.976 | 4.304 (2.0716) | 3.590 |  | 6.549 (0.5057) | 3.660 (1.2265) | 2.955 (0.9418) | 3.574 (1.7284) | 3.442 (1.4747) | 2.687 (0.8776) | 2.579 (0.3859) | 2.678 (0.7295) | 3.186 (2.2441) | 2.521 | 3.463 (0.7562) | 2.465 (0.8425)
  Day 5: number analyzed (Participants) | 6 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 1 | 0 | 9 | 2 | 5 | 6 | 6 | 7 | 6 | 3 | 5 | 1 | 5 | 2
  Day 5 | 6.604 (0.4842) | 4.578 (0.6202) | 2.581 (1.0972) | 1.748 (0.0110) | 2.996 (0.4644) |  | 2.605 | 2.689 (0.5473) | 3.117 | 4.620 (1.9568) | 3.742 |  | 6.450 (0.6437) | 4.705 (1.4275) | 3.127 (1.1484) | 3.865 (1.8868) | 3.532 (1.5350) | 2.699 (1.0083) | 2.443 (0.3787) | 2.673 (0.2813) | 3.372 (2.0433) | 2.577 | 4.123 (1.1255) | 2.907 (0.7850)
  Day 6: number analyzed (Participants) | 6 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 1 | 0 | 9 | 2 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 1 | 5 | 2
  Day 6 | 6.595 (0.3266) | 5.388 (0.5909) | 2.740 (1.2380) | 2.134 (0.3192) | 3.138 (0.5754) |  | 2.801 | 2.668 (0.7974) | 3.813 | 5.035 (1.9842) | 3.653 |  | 6.426 (0.6525) | 5.403 (1.0383) | 3.669 (1.3910) | 4.295 (1.9510) | 3.947 (1.4771) | 3.104 (1.2373) | 2.334 (0.3139) | 2.629 (0.6604) | 3.741 (1.8125) | 2.907 | 4.609 (1.2620) | 3.491 (0.8264)
  Day 7: number analyzed (Participants) | 6 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 1 | 0 | 9 | 2 | 5 | 6 | 6 | 5 | 6 | 5 | 5 | 1 | 5 | 2
  Day 7 | 6.563 (0.3311) | 5.612 (0.4912) | 3.637 (0.7489) | 2.988 (0.7310) | 3.390 (0.1908) |  | 3.312 | 2.684 (1.0300) | 4.196 | 5.038 (1.9476) | 3.713 |  | 6.504 (0.7748) | 5.604 (1.0949) | 4.276 (1.3284) | 4.704 (2.0419) | 4.449 (1.5628) | 3.862 (1.4141) | 2.034 (0.3534) | 3.034 (0.6583) | 4.394 (1.5772) | 2.877 | 5.183 (1.5012) | 3.842 (1.2488)
  Day 8: number analyzed (Participants) | 6 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 1 | 0 | 10 | 2 | 5 | 6 | 6 | 7 | 6 | 5 | 5 | 1 | 5 | 2
  Day 8 | 6.643 (0.4611) | 5.744 (0.7194) | 3.875 (0.5026) | 3.053 (1.1852) | 3.867 (0.3347) |  | 3.441 | 2.913 (1.0913) | 4.553 | 5.123 (1.6669) | 4.114 |  | 6.503 (0.5202) | 5.653 (0.8166) | 4.694 (1.3082) | 5.324 (1.8687) | 4.949 (1.4416) | 3.791 (1.5984) | 2.222 (0.4366) | 3.362 (0.7384) | 4.996 (1.4838) | 3.423 | 5.485 (1.3293) | 4.256 (1.3887)
  Day 10: number analyzed (Participants) | 5 | 2 | 3 | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 1 | 0 | 10 | 2 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 1 | 5 | 2
  Day 10 | 6.817 (0.3336) | 6.171 (0.8102) | 4.369 (0.3684) | 3.488 (1.1964) | 4.059 (0.0027) |  | 3.948 | 3.438 (1.2872) | 5.061 | 5.724 (2.0787) | 4.754 |  | 6.580 (0.5065) | 5.750 (0.5333) | 5.629 (1.5354) | 5.485 (1.6832) | 5.733 (1.5375) | 4.319 (1.6357) | 2.928 (0.8495) | 4.073 (1.1757) | 5.111 (1.2601) | 3.585 | 5.193 (0.6566) | 5.240 (1.1278)
  Day 17: number analyzed (Participants) | 6 | 2 | 3 | 1 | 2 | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 10 | 2 | 5 | 6 | 6 | 7 | 6 | 5 | 5 | 1 | 5 | 2
  Day 17 | 6.601 (0.3466) | 6.713 (0.6714) | 6.147 (1.0166) | 2.949 | 4.572 (0.1838) |  | 6.953 | 5.127 (1.8225) | 6.744 | 5.881 (1.3108) | 6.621 |  | 6.444 (0.6440) | 6.297 (0.5676) | 6.292 (0.5110) | 5.888 (1.3019) | 6.019 (0.8985) | 5.455 (1.2889) | 4.546 (1.3663) | 6.311 (1.3623) | 4.981 (0.9912) | 6.260 | 5.987 (0.6606) | 5.383 (0.8259)

8. Secondary Outcome: Pharmacokinetic (PK) Parameter of Velpatasvir: AUCinf
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: 0 (predose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose at Day 1
Population: The PK analysis set included all randomized and treated participants who have evaluable PK profiles for velpatasvir.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 4 | 15 | 12 | 8 | 30
h*ng/mL | 113.8 (71.61) | 857.9 (612.23) | 2054.3 (806.69) | 2727.3 (1619.74) | 4546.6 (1757.10)

9. Secondary Outcome: PK Parameter of Velpatasvir: AUCtau
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: 0 (predose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose at Day 3
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 4 | 15 | 12 | 8 | 30
h*ng/mL | 86.4 (14.32) | 857.5 (467.74) | 1950.5 (486.87) | 2745.3 (1480.47) | 5003.0 (2371.91)

10. Secondary Outcome: PK Parameter of Velpatasvir: Cmax
Description: Cmax is defined as the maximum observed plasma concentration of drug.
Time Frame: 0 (predose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose at Day 1 for single dose and Day 3 for multiple dose.
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 4 | 15 | 12 | 8 | 30
ng/mL
  Day 1 (Single-Dose) | 20.1 (14.62) | 110.8 (55.97) | 272.3 (95.46) | 372.8 (222.74) | 583.3 (257.90)
  Day 3 (Multiple-Dose) | 16.2 (2.34) | 122.9 (61.38) | 292.4 (88.77) | 413.9 (243.66) | 690.1 (307.04)

11. Secondary Outcome: PK Parameter of Velpatasvir: CL/F
Description: CL/F is defined as the apparent oral clearance following administration of the drug.
Time Frame: as for outcome 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 4 | 15 | 12 | 8 | 30
mL/hr
  Day 1 | 61312.2 (42726.76) | 37170.7 (16570.51) | 27930.6 (10689.18) | 49237.5 (25550.98) | 38011.7 (14392.55)
  Day 3 | 59173.6 (10490.08) | 34,820.1 (13217.45) | 27,263.0 (7367.47) | 53,194.3 (39618.97) | 37,362.8 (18382.06)

12. Secondary Outcome: PK Parameter of Velpatasvir: Ctau
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: 0 (predose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose at Day 3
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
Number analyzed (Participants) | 4 | 15 | 12 | 8 | 30
ng/mL | 0.6 (0.70) | 10.8 (8.50) | 22.4 (4.66) | 30.8 (15.03) | 60.6 (33.24)

13. Secondary Outcome: Number of Participants With Nonstructural Protein 5A (NS5A) Resistance Associated Variants (RAVs) at Pretreatment or Postbaseline Timepoints
Description: The full-length NS5A coding region was analyzed pretreatment (baseline) by deep sequencing using MiSeq for all 70 participants who received velpatasvir and for 8 of 17 participants who received placebo prior to and up to 2 weeks (Day 17) after dosing with velpatasvir. Participants were categorized by velpatasvir dose/HCV genotype and presence or absence of NS5A RAVs.
Time Frame: First dose date up to Day 17
Population: Participants in the efficacy analysis set who were sequenced at pre-treatment or post baseline treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Velpatasvir 5 mg (GT 1a) | Velpatasvir 25 mg (GT 1a) | Velpatasvir 50 mg (GT 1a) | Velpatasvir 100 mg (GT 1a) | Velpatasvir 150 mg (GT 1a) | Velpatasvir 150 mg (GT 1b) | Velpatasvir 150 mg (GT 2) | Velpatasvir 25 mg (GT 3) | Velpatasvir 50 mg (GT 3) | Velpatasvir 150 mg (GT 3) | Velpatasvir 150 mg (GT 4)
Number analyzed (Participants) | 8 | 4 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 4 | 6 | 2
Participants
  Number of participants sequenced pretreatment | 8 | 4 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 4 | 6 | 2
  Number of participants with RAVs at pretreatment | 2 | 0 | 2 | 3 | 3 | 2 | 1 | 4 | 2 | 1 | 2 | 2
  Number of participants sequenced at postbaseline | 2 | 4 | 8 | 7 | 8 | 6 | 6 | 8 | 6 | 4 | 6 | 2
  Number of participants with RAVs at postbaseline | 0 | 4 | 7 | 6 | 8 | 6 | 6 | 7 | 6 | 4 | 6 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Day 17 + 2 (Day 19 if Day 17 visit missing); All-Cause Mortality: First dose date up to Week 48
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug (velpatasvir or placebo). Data were summarized by velpatasvir and placebo.
Arm/Group | Placebo | Velpatasvir 5 mg | Velpatasvir 25 mg | Velpatasvir 50 mg | Velpatasvir 100 mg | Velpatasvir 150 mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/4 | 0/15 | 0/12 | 0/8 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/4 | 0/15 | 0/12 | 0/8 | 0/31
Other Adverse Events (participants affected / at risk) | 3/17 | 1/4 | 4/15 | 1/12 | 3/8 | 6/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Velpatasvir 5 mg (N=4) | Velpatasvir 25 mg (N=15) | Velpatasvir 50 mg (N=12) | Velpatasvir 100 mg (N=8) | Velpatasvir 150 mg (N=31)
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 4
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years